CLINICAL TRIAL: NCT05106634
Title: Evaluation of Breastfeeding Success and Self-Efficacy Using LATCH in Mothers Giving Birth Via Vaginal Delivery or Cesarean Section: Cross-sectional Study
Brief Title: Evaluation of Breastfeeding Success and Self-Efficacy in Mothers Giving Birth Via Vaginal Delivery or Cesarean Section
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Gonca Buran, RN, PhD, lecturer, Uludag University
Other Study IDs: 2019-14/18
Record Dates: First submitted 2021-10-23; First posted 2021-11-04 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2021-10

CONDITIONS: Breastfeeding
Keywords: Breastfeeding Success; breastfeeding Self-Efficacy; vaginal delivery; cesarean section; spinal anesthesia; general anesthesia; epidural anestezi
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This cross-sectional observational study was conducted to compare breastfeeding success and breastfeeding self-efficacy levels of mothers who gave birth via vaginal delivery (spontaneous or via epidural analgesia) or cesarean section (under general or spinal anesthesia).

DETAILED DESCRIPTION:
This study was conducted by including women, who gave birth via VD or CS in the gynecology clinics of a training and research hospital and a city hospital and were in the postpartum period (after 24 hours).

It compared the breastfeeding self-efficacy and breastfeeding success of mothers who gave birth via CS (under spinal anesthesia or general anesthesia) with those of mothers who gave birth via vaginal delivery (under epidural analgesia or via spontaneous vaginal delivery).

ELIGIBILITY:
Inclusion Criteria:

1. being aged >18 years old;
2. being literate;
3. having a baby of weight between 2500-4000 g, with 5th minute APGAR score of ≥7, and without congenital diseases and sucking and swallowing problems;
4. not having a disease that prevents breastfeeding;
5. having a full-term (37-42 weeks) VD or CS,
6. agreeing to participate in the study

Exclusion Criteria:

1. a history of psychological or mental health problems
2. any condition in the mother or infant that was a barrier to breastfeeding
3. baby's admission into the neonatal unit
4. baby's separation from the mother for any reason

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Being aged >18 years old women who gave birth via VD or CS in the gynecology clinics of a training and research hospital and a city hospital and were in the early postpartum period (after 24 hours)
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Breastfeeding success observing | Postpartum 24 hours
  assessed using the LATCH Breastfeeding Assessment Tool
Breastfeeding Self-Efficacy | Early postpartum period (after 24 hours)
  assessed using the Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF)

CONTACTS AND LOCATIONS:
Overall Officials: Gonca Buran, PhD, Principal Investigator — Uludag Üniversity
Locations (1):
- Ul, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alus Tokat M, Sercekus P, Yenal K, Okumus H. Early postpartum breast-feeding outcomes and breast-feeding self-efficacy in Turkish mothers undergoing vaginal birth or cesarean birth with different types of anesthesia. Int J Nurs Knowl. 2015 Apr;26(2):73-9. doi: 10.1111/2047-3095.12037. Epub 2014 Jun 5. PMID 24897921
- [Background] Maharlouei N MD, Pourhaghighi A Medical student, Raeisi Shahraki H PhD, Zohoori D MD, Lankarani KB MD. Factors Affecting Exclusive Breastfeeding, Using Adaptive LASSO Regression. Int J Community Based Nurs Midwifery. 2018 Jul;6(3):260-271. PMID 30035142